CLINICAL TRIAL: NCT03393871
Title: Myocardial Mass Determination of the Different Coronary Territories by FFRct and Invasive Measurement of Absolute Coronary Blood Flow. A Clinical Registry
Brief Title: Myocardial Mass Determination by FFRct and Absolute Coronary Blood Flow
Acronym: MyoMass
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Nico Pijls, Dr. PHD, Catharina Ziekenhuis Eindhoven
Other Study IDs: MyoMass
Record Dates: First submitted 2017-12-28; First posted 2018-01-09 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2018-02

CONDITIONS: Fractional Flow Reserve; Absolute Flow Measurement; FFR-CT; Myocardial Mass; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: absolute blood flow measurement — Absolute maximum flow will be measured, using the RayFlow® multifunctional monorail infusion catheter. (This measurement takes a few minutes per artery, does not require any additional drug, but only 50-100 ml of saline per artery, and is not associated with any additional risk for the patient compared to the regular invasive procedure.

SUMMARY:
The background for performing the present study is to compare the mass calculations by CT scanning and by invasive absolute blood flow measurements and thereby corroborating both methods.

DETAILED DESCRIPTION:
Although knowledge about the myocardial mass (in grams) of the different territories belonging to the major coronary arteries, is of clinical importance to estimate risk of coronary interventions (PCI, CABG) and to determine area of necrosis after myocardial infarction, no invasive methodology has been available so far for reliable assessment of mass.

Especially in the setting of percutaneous coronary intervention (PCI), it would be valuable to have information about the absolute and relative myocardial mass distal to the location where the intervention is planned. Such information is valuable for risk estimation and can also be helpful in multivessel disease to determine the most adequate way of revascularization.

Both MRI and CT scanning have claimed to be able to estimate myocardial mass non-invasively, but by the lack of any gold standard, none of these methods could be validated in vivo so far.

A relatively new development in CT technology is the calculation of fractional flow reserve (FFR) by CT scanning, according to a sophisticated algorithm developed by Heartflow Inc. One of the baseline assumptions in that algorithm is that myocardial mass is proportional to resting blood flow, which seems a plausible assumption from a rational physiological point of view.

More recently, invasive calculation of absolute blood flow has become possible as well as resistance measurement of the (microcirculation of the) myocardium.

Using that invasive technology (explained in the appendix to this protocol), it can be assumed that measuring absolute maximum blood flow in a coronary artery as well as fractional flow reserve for different territories or for different spots within one major coronary artery, provides a basis for relative mass calculation. The background for performing the present study is to compare these mass calculations by CT scanning and by invasive measurements, thereby corroborating both methods.

ELIGIBILITY:
Inclusion Criteria:

* Presence of multivessel coronary disease with an indication for multivessel FFR and/or PCI or patients with single vessel disease scheduled for FFR/PCI of that single coronary artery
* Availability of a coronary CT scan performed prior to the scheduled invasive investigation. The time difference between the CT scan and the invasive exam should be less than 3 months.
* Focal lesions only
* Normal left ventricular function
* Age < 75 years
* Note: previous uncomplicated PCI in any of the coronary arteries is permitted

Exclusion Criteria:

* Inability to give informed consent
* Diffuse coronary disease
* Tortuous or calcified arteries interfering with reliable invasive FFR assessment
* Previous myocardial infarction or ejection fraction less than 60% by echocardiography or ventriculography or less than 50% by nuclear methods
* Atrial fibrillation interfering with high quality coronary CT scanning
* Contra-indications for CT scanning
* Left main stenosis
* Age > 75 years
* Pregnancy or desired pregnancy in the future

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients will be included who are scheduled
  1. Either for multivessel FFR/PCI fulfilling the following criteria and not meeting any of the exclusion criteria (prospective group)
  2. Or patients in whom both coronary CT scanning and invasive exams have been performed already for clinical reasons and of whom "complete data" are available already (retrospective group)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Mass and flow | 3 months
  To compare relative myocardial mass distribution (i.e. mass of the respective territories of LAD, LCX and RCA) by CT scanning to normalized hyperemic blood flow in the three major myocardial territories as assessed by absolute flow measurements and FFR in patients with an indication for multivessel FFR measurement.
Comparison of Mass and flow in the LAD | 3 months
  To compare relative myocardial mass belonging to a proximal or a mid segment of one of the major coronary arteries measured by CT scanning to invasive absolute flow and FFR measurement in that particular proximal or mid coronary artery in patients undergoing single or multivessel PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Nico HJ Pijls, MD, PhD, Study Director — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided